CLINICAL TRIAL: NCT04145739
Title: The Sequelae of Mastectomy and Quadrantectomy Respect to the Reaching Movement in Breast Cancer Survivors: the Evidences of an Integrated Rehabilitation Protocol During the Oncological Care Path
Brief Title: The Sequelae of Mastectomy and Quadrantectomy Respect to the Reaching Movement in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Teresa Paolucci, Medical Doctor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URomLS-2019
Record Dates: First submitted 2019-10-23; First posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer; Pain, Chronic; Pain, Postoperative; Mastectomy; Lymphedema
Keywords: Breast Cancer; Pain, Chronic and Postoperative; Posture; Target - Reaching movement; Mastectomy; Quadrantectomy; Lymphedema; Rehabilitation; Scapula tilting; Shoulder; Biomechanics; Upper limb
MeSH Terms: conditions — Breast Neoplasms; Chronic Pain; Pain, Postoperative; Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mastectomy group (Experimental): Patients undergoing mastectomy
  Interventions: Other: Rehabilitation protocol
- Quadrantectomy group (Experimental): Patients undergoing quadrantectomy
  Interventions: Other: Rehabilitation protocol

INTERVENTIONS:
Other: Rehabilitation protocol — The rehabilitation treatment was performer in single session, lasted 60 minutes for session, 2 times a week, carried-out a 6-week exercises program for a total of 12 sessions, by a physiotherapist trained in oncologic rehabilitation, who started with a first phase of at least 15-20 min of low-impact aerobics warm-up. The second phase consisted in diaphragmatic breathing and postural exercises for the midline alignment in a supine position. Finally the patient continued in front of the mirror with exercises for the recovery of shoulder joint, isometric reinforcement exercises for the recovery of strength of shoulder stabilizer muscles. In the presence of lymphedema an additional weekly lymph drainage session was performed for a total of 10 sessions.

SUMMARY:
The hypothesis behind our study was that patients after BC surgery, who underwent quadrantectomy or mastectomy, may present a different disability respect to the upper limb on the operated side. Accordingly they could have a different functional recovery patterns after rehabilitation.

The aim of our study was to compare the recovery of the fluidity of the reaching movement (Jerk) as the primary outcome, the reduction of shoulder pain and improvement of disability for the upper limb respect the operated side as secondary outcomes, before and after a specific rehabilitation protocol treatment.

DETAILED DESCRIPTION:
Surgery is usually the first line of attack against breast cancer (BC). The decisions about surgery depend on many factors based on the stage, the type of cancer and patient acceptability, in terms of her long term peace of mind and survival prospects. Typically, breast reconstruction takes place during or soon after mastectomy, to avoid psychological distress for the patient, and in some cases, also after lumpectomy or quadrantectomy; furthermore breast reconstruction can be done many months or even years after surgery too.

Today, breast cancer rehabilitation can help survivors to obtain and maintain the highest possible physical, social, psychological and vocational functioning, within the limits created by cancer and its treatments. After BC surgery, is common to detect disorders as shoulder dysfunction, postmastectomy syndrome, chemotherapy-induced peripheral neuropathy, axillary cording, lymphedema and a host of others as postural imbalance.

Also, alterations in muscle activation and restricted shoulder mobility, which are common in BC patients, have been found to affect upper limb function and alterations in muscle activity patterns differed by breast surgery and reconstruction type: rehabilitation and in particular mobilization stretches and shoulder and scapula exercises after breast surgery are an effective resource to improve upper limb range of motion and decrease chest tightness and pain.

This study was prompted by the lack of literature about the quadrantectomy versus mastectomy intervention, considering the disability of the upper limb from the operated side, especially if in relation to the rehabilitation pathway, currently recommended in BC care.

ELIGIBILITY:
Inclusion Criteria:

* total mastectomy with breast prostheses or tissue expanders performed or quadrantectomy
* age from 18 to 60 years
* body mass index (BMI) < 30
* no cognitive dysfunctions ( Mini Mental State Examination MMSE > 24)
* mild lymphedema

Exclusion Criteria:

* presence of lymphangitis or mastitis
* presence of metastasis
* surgical complications of the intervention, neurological deficits and complications
* important shoulder joint problems before the intervention for BC
* severe-moderate lymphedema and web axillary syndrome
* visual problem not corrected by lenses
* other or previous physiotherapy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Time variation of the normalized jerk (NJ) within biomechanical reaching movement | T0 baseline - T1 (30 days) - T2 (3 months)
  The normalized jerk (NJ) was evaluated through the Smart D500 stereo-photogrammetric system (BTS, Italy), calculated on the wrist-target marker distance, within the reaching task performed on the side underwent surgery. It measures the fluidity of the upper limb movement.

SECONDARY OUTCOMES:
Time variation of Visual Analogue Scale (VAS) | T0 baseline - T1 (30 days) - T2 (3 months)
  Instrument to assess unidimensional measure of pain intensity. VAS was presented in a coloured scale with a middle point, graduations and numbers. Under the scale there was a straight horizontal line of fixed length, 100 mm. The ends were defined as the limits of the parameter to be measured (pain in the last 24 hours), orientated from the left (worst, no pain) to the right (best, worst pain to be imagined). The score is determined by measuring the distance (cm) on the 10 cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-10.
Time variation of Disabilities of Arm, Shoulder and Hand Questionnaire (DASH) | T0 baseline - T1 (30 days) - T2 (3 months)
  Self-administered region-specific outcome instrument developed as a measure of self-rated upper-limb disability and symptoms, actually used to monitor changes in symptoms and function over time. It consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100. The items are related to the degree of difficulty in performing various functional activities because of arm, shoulder or hand limitations (21 items), the intensity of pain, activity-related pain, tingling, weakness and stiffness (5 items), and the effect related to social activities, job, sleep and its psychological impact (4 items).
Time variation of Movement Duration (MD) of biomechanical reaching movement | T0 baseline - T1 (30 days) - T2 (3 months)
  The movement duration (MD) was evaluated in seconds, through the Smart D500 stereo-photogrammetric system (BTS, Italy), within the reaching task performed on the side underwent surgery.
Time variation of the angle of arm flexion at end of movement (AAF) within biomechanical reaching movement | T0 baseline - T1 (30 days) - T2 (3 months)
  The degrees of the angle of arm flexion at end of movement (AAF) were evaluated through the Smart D500 stereo-photogrammetric system (BTS, Italy), within the reaching task performed on the side underwent surgery. A zero value is conventionally assigned to AAF when the arm is along the side, positive values represent flexion, negative ones represent extension.
Time variation of the angle at elbow at end of movement (AE) within biomechanical reaching movement | T0 baseline - T1 (30 days) - T2 (3 months)
  The degrees of the angle at elbow at end of movement (AE) were evaluated through the Smart D500 stereo-photogrammetric system (BTS, Italy), within the reaching task performed on the side underwent surgery. The value assigned is zero when the elbow is completely extended, positive values correspond to flexion, and negative ones to hyperextension.
Time variation of the mean value of target-approaching velocity (TAV) within biomechanical reaching movement | T0 baseline - T1 (30 days) - T2 (3 months)
  The mean value of target-approaching velocity (TAV) was evaluated through the Smart D500 stereo-photogrammetric system (BTS, Italy), within the reaching task performed on the side underwent surgery.

OTHER OUTCOMES:
Time variation of range of Motion (ROM) of shoulder | T0 baseline - T1 (30 days) - T2 (3 months)
  The degrees of flexion, extension, adduction, abduction and internal and external rotation evaluated on the side underwent surgery.
Time variation of muscular strength regards shoulder ROM | T0 baseline - T1 (30 days) - T2 (3 months)
  Parameters evaluated according to the scale of Medical Research Council Manual Muscle Testing (MRC), on a scale of 0 to 5 in relation to the maximum expected for that muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Paolucci, MD, PhD, Principal Investigator — University 'Sapienza' of Rome
Locations (1):
- Umberto I Hospital, Rome, Italy